CLINICAL TRIAL: NCT03338764
Title: A Double-Blind, Placebo-Controlled, Parallel Design Phase 3 Study to Assess the Efficacy, Safety, Tolerability, and Pattern of Use of SM-1 in Adult Subjects With a History of Transient Insomnia
Brief Title: An Investigational Study to Assess Efficacy and Pattern of Use of SM-1 in Subjects With a History of Transient Insomnia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Sequential Medicine Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SM-A-06
Record Dates: First submitted 2017-11-03; First posted 2017-11-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Transient Insomnia
Keywords: Transient insomnia; Insomnia; Sleep initiation and maintenance disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (SM-1) (Experimental): Drug: SM-1 3-drug combination product containing 50-mg diphenhydramine, 5-mg delayed-release zolpidem and 0.5-mg delayed-release lorazepam.
  Interventions: Drug: SM-1
- Placebo (Placebo Comparator): Drug: Placebo Identical in appearance to SM-1 and has the same excipients, but no active ingredients or delayed-release coating materials.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SM-1 — SM-1 3-drug combination product containing 50-mg diphenhydramine, 5-mg delayed-release zolpidem and 0.5-mg delayed-release lorazepam self-administered as needed to promote sleep
  Arms: Experimental (SM-1)
Drug: Placebo — Identical in appearance to SM-1 and has the same excipients, but no active ingredients or delayed-release coating materials, self-administered as needed to promote sleep
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and pattern of use of the combination drug product SM-1 in adults who sometimes have difficulty in falling asleep or staying asleep, but who do not have chronic insomnia. Participants will receive SM-1 or placebo to take at home as needed over the course of 3 months treatment period.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy, safety, tolerability and pattern of use of SM-1 in adults who sometimes have difficulty in falling asleep or staying asleep, but who do not have chronic insomnia. SM-1 is a combination drug product containing diphenhydramine, zolpidem and lorazepam. The study is a parallel group design; participants will receive either SM-1 or placebo to take at home as needed over the course of 3 months treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Experienced at least 1 prior episode of transient insomnia meeting all of the following criteria: difficulty falling asleep or staying asleep; next day impairment or distress associated with the disturbed sleep; frequency of 1 to 7 nights per week; duration of less than 1 month or more than 1 month of intermittent episodes.
* Routinely spends 6.5 - 9.5 hours in bed each night, with bed time varying no more than 2 hours over a week.
* Body Mass Index (BMI) between 19 and 32 kg/m2.
* Good general health, as determined by a thorough medical, sleep and psychiatric history review, brief physical examination including vital sign measurements, and an assessment of screening laboratory test results.
* Agrees, for the duration of the study, to take only study drug to address difficulty falling asleep or staying asleep, and to not drink alcohol within 2 hours of expected bedtime.

Exclusion Criteria:

* Females who are pregnant, breast-feeding, or planning a pregnancy during the study period.
* Clinically significant medical disorder or currently unstable medical condition that, in the opinion of the investigator, would confound the results of the study.
* Abnormal laboratory value at screening, judged clinically significant by the investigator.
* History or current evidence of severe hepatic (liver) impairment.
* Clinically significant psychiatric illness, or the history or presence of a major psychiatric illness in the past year.
* Has a significant risk (in the opinion of the investigator) for suicidal behavior during the course of participation in the study or a) At screening: the subject scores "yes" on items 4 or 5 in the Suicidal Ideation section of the C-SSRS with reference to a 6-month period prior to screening; or b) At screening: the subject has had one or more suicidal attempts within a 2-year period prior to screening; or c) At the baseline visit: the subject scores "yes" on items 4 or 5 in the Suicidal Ideation section of the C-SSRS with reference to screening; or d) The subject is considered to be an imminent danger to self or others.
* Has a history of chronic insomnia or other sleep disorders, such as sleep apnea, narcolepsy, parasomnia, restless leg syndrome, or circadian rhythm disorder.
* Has used medications to aid sleep on most nights during the past 2 months.
* Has a history of night work or shift work within the month prior to screening or a need to participate in night work or shift work during the study.
* Has a history of alcohol or substance use disorder within the year prior to screening, or current evidence of alcohol or substance use disorder as defined by the Diagnostic and Statistical Manual of the American Psychiatric Association, 5th Edition.
* Self-report of a usual consumption of more than 14 units of alcohol per week: 1 unit of alcohol is equivalent to 12 ounces of beer, 4 ounces of wine, or 1 ounce of liquor.
* Has a history of routinely smoking during sleep period.
* Has discontinued smoking or participated in a smoking cessation program within 28 days of screening, or plans to discontinue smoking during the study.
* Has used within 2 weeks or 5 half-lives (whichever is longer) prior to screening of any medication that affects sleep-wake function.
* Has a positive urine drug screen at the screening visit.
* Has a history of allergy or known sensitivity, hypersensitivity, or adverse reaction to diphenhydramine, zolpidem, lorazepam, or related compounds.
* Has had treatment with any other investigational drug within 28 days or 5 half-lives (whichever is longer) prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Subjective Total Sleep Time | 7 nights
  Total time spent sleeping each night as reported by the subject

SECONDARY OUTCOMES:
Pattern of use | 3 months
  Subject reported total number of uses and consecutive nights of use
Safety Adverse Events | Through study completion, 17 weeks
  Adverse Events
Safety Residual Effects | Through study completion, 17 weeks
  Subject reported answer to the Question, "How alert or sleepy do you feel this morning?" Subjects will rate their alertness on a scale from 0 to 5, with 0 being extremely sleepy and 5 being extremely alert
Safety Rebound Insomnia | Through study completion, 17 weeks
  Total time spent sleeping each night as reported by the subject on night after taking drug or night after not taking drug